CLINICAL TRIAL: NCT06491251
Title: Outcomes of Varicocelectomy in Patients With Clinical Varicocele and Unexplained Infertility
Brief Title: Varicocelectomy in Patients With Clinical Varicocele and Unexplained Infertility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Abd El-Moaty Khalifa, Principle Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unexplained male infertility
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Unexplained Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varicocelectomy group (Experimental): Bilateral Subinguinal microscopic varicocelectomy
  Interventions: Procedure: Bilateral Subinguinal microscopic varicocelectomy
- Controlled group (No Intervention): no intervention , follow up

INTERVENTIONS:
Procedure: Bilateral Subinguinal microscopic varicocelectomy — Using Leica® Microsystems , Germany. the patient was placed in a supine position after spinal anesthesia administration , The left external inguinal ring was located near the pubic tubercle by palpation, and the incision site was marked below the annulus of the left external ring. A 1.5- to 3-cm oblique incision was made along the skin line. After the tissues were dissected layer by layer, the incision was exposed until the spermatic cord became visible. the spermatic cord was lifted out with Babcock clamp and delivered though the incision and followed by the placement of a nelaton catheter 20 fr below the spermatic cord. The external spermatic vein was located and ligated. The microscopic operation was performed at 10× to 20× magnification.
  Arms: Varicocelectomy group

SUMMARY:
This study was conducted to assess the efficacy of varicocelectomy in unexplained male infertility with clinical varicocele The primary objective was to assess the pregnancy outcomes in these group. The secondary objective was to analyses improvement in Sperm DNA fragmentation , hormonal profile and semen parameter after varicocelectomy in Unexplained infertility .

DETAILED DESCRIPTION:
Infertility is defined as the absence of a desired pregnancy following regular, unprotected sexual intercourse for a period of at least 1 year. Over 15% of married couples worldwide experience fertility problems, and 50% of these cases are caused by male factor infertility.

Varicocele is the abnormal enlargement of the veins within the pampiniform plexus. The condition affects approximately 15% of the overall adult male population and 35% of men with primary infertility. Among men with secondary infertility, varicose veins are found in up to 80% of patients.

Only about 20% of all men with varicocele present with infertility. But overall, it is the most frequent abnormality found in infertile men.

Microsurgical varicocelectomy has gradually become the preferred surgical option for varicocele due to its advantages of less surgical damage, lower postoperative recurrence rate, fewer complications, higher postoperative semen quality, and higher postoperative fertility rate.

The two approaches to microsurgical varicocelectomy include the inguinal or subinguinal routes. The subinguinal approach involves the shallow spermatic cord and simple anatomic layers; it does not require the dissection of the external abdominal oblique muscle and allows for the application of spinal anesthesia.

Sub-inguinal approach assisted by microscope magnification is a safe, simple , and effective method for the treatment of sub fertile men and permit significant improvement in DNA fragmentation index and sperm parameters.

Varicocele is linked to male infertility through various nonmanually exclusive mechanisms, including an increase in the production of reactive oxygen species (ROS) that may lead to sperm deoxyribonucleic acid (DNA) damage.

Excessive sperm DNA breaks, so-called sperm DNA fragmentation (SDF), are commonly found in the ejaculates of men with varicocele and fertility-related issues. Although elevated SDF is mainly observed in men with abnormal semen parameters, namely, count, motility, and morphology, it can coexist with normozoospermia.

Semen analysis is the most important test for evaluating male infertility, but it does not provide information regarding all functions of sperm, nor is it sufficient for predicting male fertility potential and the likelihood of success of assisted reproductive technology (ART).

Furthermore, the standards for normal values in semen analysis do not reflect average values, In fact, 15% of patients with male infertility were found to have normal semen analysis results. Therefore, additional tests should be performed due to the limitations of using semen analysis results alone to evaluate male fertility potential.

Sperm DNA fragmentation (SDF) testing measures the quality of sperm as a DNA package carrier, and it therefore is more significant than the parameters analyzed in previous semen analyses.

Elevated SDF was shown to impair natural fertility and assisted reproductive (ART) outcomes.

SDF can be observed even in men with normal semen analysis results. Damage to sperm DNA can result in longer time to pregnancy, unexplained infertility, recurrent pregnancy loss, Therefore, interventions aimed at explored to potentially improve natural fertility.

This study was conducted to assess the efficacy of varicocelectomy in unexplained male infertility with clinical varicocele The primary objective was to assess the pregnancy outcomes in these group. The secondary objective was to analyses improvement in Sperm DNA fragmentation , hormonal profile and semen parameter after varicocelectomy in Unexplained infertility .

ELIGIBILITY:
Inclusion Criteria:

* Patients unable to conceive after 12 month of regular and unprotected intercourse
* Male patients aged 18 -45 years old
* Normal semen analysis (concentration, motility and morphology) according to WHO criteria 2021
* Infertile men with clinical varicocele (grade II,III) subjected to varicocelectomy
* No history of other congenital or acquired urogenital diseases
* Primary infertility
* Normal BMI (18.5-24..9)

Exclusion Criteria:

* History of other congenital or acquired urogenital diseases
* Age outside inclusion criteria
* Grade I varicocele confirmed by ultrasound ( subclinical varicocele )
* Abnormal semen analysis
* Recurrent varicocele
* Patient unable or unwilling to comply with follow-up schedule
* Female fertility issues (anovulation , hormonal infertility, tubal factor, endometriosis)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
varicocelectomy improved spontaneous pregnancy rates | follow up 1 year post varicocelectomy
  Sub inguinal microscopic varicocelectomy increase spontaneous pregnancy rates in groups with high sperm DNA fragmentation index in comparison to control group or varicocelectomy group with intermediate or normal sperm DNA fragmentation index
Effect of Infertility duration on sperm parameter and pregnancy rate after varicocelectomy | follow up 1 year post varicocelectomy
  The infertility duration is sub grouped into three according to months of primary infertility and measures changes in sperm concentration , motility ,morphology and changes in spontaneous pregnancy rate in different groups

SECONDARY OUTCOMES:
Improvement in Sperm DNA fragmentation index | follow up 1 year post varicocelectomy
  decrease of sperm DNA fragmentation index after varicocelectomy in group with high sperm DNA fragmentation index > 25 %
Changes in sperm concentration , Motility and morphology after varicocelectomy | follow up 1 year post varicocelectomy
  increasing in sperm concentration , Motility and morphology after varicocelectomy in group with High sperm DNA fragmentation index > 25% in comparison to group with normal sperm DNA fragmentation index

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Khalifa, MSc, Principal Investigator — Kafrelsheikh University; Tarek M. Abdelbaky, MD, Study Director — Kafrelsheikh University; Ayman S. Rashed, MD, Study Director — October 6 University; Khaled M. Magdy Zeinelabden, MD, Study Director — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Egypt

REFERENCES:
- [Background] Dai Y, Liu J, Yuan E, Li Y, Shi Y, Zhang L. Relationship Among Traditional Semen Parameters, Sperm DNA Fragmentation, and Unexplained Recurrent Miscarriage: A Systematic Review and Meta-Analysis. Front Endocrinol (Lausanne). 2022 Jan 4;12:802632. doi: 10.3389/fendo.2021.802632. eCollection 2021. PMID 35058886
- [Background] Guzick DS, Overstreet JW, Factor-Litvak P, Brazil CK, Nakajima ST, Coutifaris C, Carson SA, Cisneros P, Steinkampf MP, Hill JA, Xu D, Vogel DL; National Cooperative Reproductive Medicine Network. Sperm morphology, motility, and concentration in fertile and infertile men. N Engl J Med. 2001 Nov 8;345(19):1388-93. doi: 10.1056/NEJMoa003005. PMID 11794171